CLINICAL TRIAL: NCT05070858
Title: Efficacy and Safety of Pozelimab and Cemdisiran Combination Therapy and Cemdisiran Monotherapy in Patients With Symptomatic Generalized Myasthenia Gravis
Brief Title: A Study to Test How Safe Pozelimab and Cemdisiran Combination Therapy and Cemdisiran Alone Are and How Well They Work in Adult Patients With Generalized Myasthenia Gravis
Acronym: NIMBLE
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R3918-MG-2018; 2020-003272-41 (EudraCT Number); 2023-508842-17-00 (EU CTIS Number)
Record Dates: First submitted 2021-09-27; First posted 2021-10-07 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Generalized Myasthenia Gravis
MeSH Terms: conditions — Myasthenia Gravis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group 1 (Experimental): Placebo in DBTP; Re-randomized to Combination or Cemdisiran in ETP and OLTP
  Interventions: Drug: Pozelimab + Cemdisiran; Drug: Cemdisiran; Other: Placebo
- Group 2 (Experimental): Combination regimen throughout the study. For participants who have not reached week 108 will receive cemdisiran monotherapy in the OLTP.
  Interventions: Drug: Pozelimab + Cemdisiran; Drug: Cemdisiran
- Group 3 (Experimental): Cemdisiran throughout the study
  Interventions: Drug: Cemdisiran
- Group 4 (Experimental): Pozelimab monotherapy in DBTP followed by combination in ETP and OLTP. For participants who have not reached week 108 will receive cemdisiran monotherapy in the OLTP.
  Interventions: Drug: Pozelimab + Cemdisiran; Drug: Cemdisiran; Drug: Pozelimab

INTERVENTIONS:
Drug: Pozelimab + Cemdisiran — Subcutaneous administration as described in the protocol
  Arms: Group 1; Group 2; Group 4
Drug: Cemdisiran — SC administration as described in the protocol
  Other Names: ALN-CC5
Other: Placebo — SC administration as described in the protocol
  Arms: Group 1
Drug: Pozelimab — SC administration as described in the protocol
  Other Names: REGN3918
  Arms: Group 4

SUMMARY:
This study is researching the experimental drugs called pozelimab and cemdisiran, and cemdisiran monotherapy. The study is focused on patients with generalized Myasthenia Gravis (gMG). Myasthenia gravis is a disease that causes weakness and fatigue in muscles in the body because the nerves and muscles are not communicating properly.

The aim of the study is to see how effective pozelimab and cemdisiran are when used in combination and when pozelimab and cemdisiran are used alone for patients with gMG.

The study is looking at several other research questions, including:

* What side effects may happen from taking the study drugs
* How the study drugs work inside the body
* How much of the study drugs are in the blood at different times
* Whether the body makes antibodies against pozelimab and cemdisiran (which could make the drugs less effective or could lead to side effects)

DETAILED DESCRIPTION:
DBTP- Double Blind Treatment Period (24 weeks) ETP - Extension Treatment Period (28 weeks) OLTP- Open Label Treatment Period (68 weeks) FUP-Off treatment Follow Up Period (52 weeks)

ELIGIBILITY:
Key Inclusion Criteria:

1. Male or female participants ≥18 years of age at screening (or ≥ legal age of adulthood based on local regulations, whichever is older)
2. Participant with documented diagnosis of Myasthenia Gravis (MG) based on medical history and supported by previous evaluations as described in the protocol
3. Documented prior history of positive serologic test or a positive result during screening of Anti-acetylcholine Receptor (AChR) antibodies or anti-Lipoprotein Receptor-related Protein 4 (LRP4) antibodies.
4. Myasthenia Gravis Foundation of America (MGFA) Clinical Classification Class II to IVa at screening
5. Myasthenia Gravis-Activities of Daily Living (MG-ADL) score ≥6 at screening. Ocular items should not contribute more than 50% of MG-ADL total score as described in the protocol
6. Currently receiving an acetylcholinesterase inhibitor or documented reason for not using acetylcholinesterase inhibitor therapy per investigator
7. Currently receiving an Immunosuppressive Therapy (IST) for MG, or documented reason why the participant is not taking an IST per investigator
8. If currently receiving an IST, not anticipated to have IST dosage changed before randomization or during Double-Blind Treatment Period (DBTP).
9. Willing and able to comply with clinic visits and study-related procedures, including completion of the primary series of the meningococcal vaccinations required per protocol

Key Exclusion Criteria:

1. Patients with antibody profile that is only positive for Muscle-Specific tyrosine Kinase (MuSK) (MuSK positivity is based on a documented prior history of positive serologic test for antibodies to MuSK or a positive result during screening
2. History of thymectomy within 12 months prior to screening or planned during the study
3. History of malignant thymoma (patients with stage 1 may be enrolled), or history of cancer within the past 5 years, except for adequately treated basal cell skin cancer, squamous cell skin cancer, or in situ cervical cancer
4. Myasthenic crisis or MGFA Class V within 1 month of screening
5. Not meeting meningococcal vaccination requirements and, at a minimum, documentation of quadrivalent meningococcal vaccination within 5 years prior to randomization and serotype B vaccine (when available) within 3 years prior to randomization as described in the protocol
6. Known contraindication to meningococcal vaccines (group ACWY conjugate and group B vaccines) as described in the protocol
7. Participants who require antibiotics for meningococcal prophylaxis and have a contraindication, warning, or precaution precluding the use of penicillin class and penicillin-alternative antibiotics planned to be used for prophylaxis, or a history of intolerance leading to the discontinuation of these antibiotics
8. Positive hepatitis B surface antigen or hepatitis C virus Ribonucleic Acid (RNA) during screening. NOTE: Cases with unclear interpretation should be discussed with the medical monitor
9. History of Human Immunodeficiency Virus (HIV) infection or a positive test at screening per local requirements

NOTE: Other protocol-defined Inclusion/ Exclusion Criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Actual)
Dates: Start 2021-12-14 (Actual); Primary Completion 2025-07-08 (Actual); Study Completion 2028-11-11 (Estimated)

PRIMARY OUTCOMES:
Change in Myasthenia Gravis-Activities of Daily Living (MG-ADL) total score | From baseline to week 24
  The total MG-ADL score ranges from 0 to 24 points, with higher scores indicating greater functional impairment and disability

SECONDARY OUTCOMES:
Change from baseline in Quantitative Myasthenia Gravis (QMG) score | Week 24
  QMG total scores range from 0 to 39, with higher scores representing greater impairment
Achievement of a ≥3-point reduction (improvement) in MG-ADL total score | From baseline to week 24
Achievement of a ≥5-point reduction (improvement) in QMG total score | From baseline to week 24
Achievement of a consistent response on the MG-ADL | From baseline to week 24
  A participant with a ≥2-point reduction (improvement) in MG-ADL total score on 2 or more consecutive assessments spanning 4 or more weeks during the DBTP
Achievement of Minimal Symptom Expression (MSE) | Week 24
  Score of 0 to 1 on the MG-ADL
Change from baseline in the Myasthenia Gravis Composite (MGC) total score | Week 24
  MGC score ranges from 0 to 50, with higher score indicating higher impairment
Change from baseline in Myasthenia Gravis Quality of Life (MG-QOL15r) total score | Week 24
  Total score ranges from 0 to 30 points; a higher score represents greater impairment
Achievement of a ≥2-, 4-, 5-, 6-, 7-, 8-, 9-, or 10-point reduction on MG-ADL total score | From baseline to week 24
Achievement of a ≥3-, 4-, 6-, 7-, 8-, 9-, or 10-point reduction on QMG | From baseline to week 24
Incidence and severity of Treatment-Emergent Adverse Events (TEAEs) in participants treated with pozelimab + cemdisiran, cemdisiran monotherapy or placebo | Through week 24
Incidence and severity of Serious Adverse Events (SAEs) in participants treated with pozelimab + cemdisiran, cemdisiran monotherapy or placebo | Through week 24
Incidence and severity of Adverse Events of Special Interest (AESIs) in participants treated with pozelimab + cemdisiran, cemdisiran monotherapy or placebo | Through week 24
Concentrations of total pozelimab in serum | Through study duration, approximate 172 weeks
Concentrations of total Complement component 5 (C5) in plasma | Through study duration, approximate 172 weeks
Concentrations of cemdisiran and its metabolites in plasma | Through study duration, approximate 172 weeks
Incidence of treatment-emergent Anti-Drug Antibodies (ADAs) to pozelimab over time | Through study duration, approximately 172 weeks
Incidence of treatment-emergent ADAs to cemdisiran over time | Through study duration, approximate 172 weeks
Change in total complement hemolysis activity assay (CH50) over time | Through study duration, approximately 172 weeks
Percent change in CH50 over time | Through study duration, approximately 172 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (116):
- United States (19):
  - HonorHealth Neurology 2018, Scottsdale, Arizona
  - University of California Irvine, Irvine, California
  - University of Southern California, Los Angeles, California
  - Colorado Springs Neurological Associates, Colorado Springs, Colorado
  - SFM Clinical Research, LLC, Boca Raton, Florida
  - Diverse Clinical Research, Miami, Florida
  - Aqualane Clinical Research, Naples, Florida
  - Neurological Services of Orlando, Orlando, Florida
  - Medsol Clinical Research Center Inc, Port Charlotte, Florida
  - University of South Florida Morsani Center for Advanced Healthcare, Tampa, Florida
  - NorthShore University Health System, Glenview, Illinois
  - St. Elizabeth's Hospital, O'Fallon, Illinois
  - Northwest Neurology Ltd. - Clinedge - PPDS, Rolling Meadows, Illinois
  - Wayne State University School of Medicine, Detroit, Michigan
  - Dayton Center for Neurological Disorders, Centerville, Ohio
  - University of Cincinnati Gardner Neuroscience Institute, Cincinnati, Ohio
  - Penn Medicine University City, Philadelphia, Pennsylvania
  - National Neuromuscular Research Institute, Austin, Texas
  - Nerve and Muscle Center of Texas, Houston, Texas
- Belgium (2):
  - Universitair Ziekenhuis Antwerpen, Edegem, Antwerp
  - AZ Sint-Lucas, Ghent, Oost-Vlaanderen
- Brazil (5):
  - IMV Pesquisa Neurologica, Porto Alegre, Rio Grande do Sul
  - Jordy Sinapse Medicina LTDA, Itapevi, São Paulo
  - Faculdade de Medicina Do ABC, Santo André, São Paulo
  - Pseg Centro de Pesquisa Clinica S.A, São Paulo
  - Hospital das Clinicas da Faculdade de Medicina da Universidade de Sao Paulo, São Paulo
- Canada (3):
  - University of Alberta, Edmonton, Alberta
  - London Health Sciences Centre, London, Ontario
  - Toronto General Hospital, Toronto, Ontario
- China (15):
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Guangdong Hospital of Traditional Chinese Medicine, Guangdong, Guangdong
  - Nanfang Hospital Southern Medical University, Guangzhou, Guangdong
  - The University of Hong Kong-Shenzhen Hospital, Shenzhen, Guangdong
  - The First Affiliated Hospital of Guangzhou University of Chinese Medicine, Guangzhou, Guangzhou
  - Hainan General Hospital, Haikou, Hainan
  - Renmin Hospital of Wuhan University - Hubei Provincial People's Hospital, Wuhan, Hubei
  - Xiangya Hospital Central South University, Changsha, Hunan
  - The First Hospital of Jilin University, Changchun, Jilin
  - Qilu Hospital of Shandong University (Qingdan), Qingdao, Shandong
  - Huashan Hospital Fudan University, Shanghai, Shanghai Municipality
  - The Second Affiliated Hospital of the Chinese Peoples' Liberation Army Air Force Medical University, Xi’an, Shanxi
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
- Denmark (4):
  - Aalborg Universitetshospital, Aalborg, North Denmark
  - Aarhus University Hospital, Aarhus N
  - Rigshospitalet, Copenhagen, Copenhagen
  - Odense Universitetshospital, Odense
- France (4):
  - Centre Hospitalier Universitaire de Nice, Nice, Alpes Maritimes
  - CHU Bicetre, Le Kremlin-Bicêtre
  - Centre Hospitalier Regional Universitaire (CHRU) de Nancy, Nancy
  - Hopital de la Pitie Salpetriere, Paris
- Georgia (5):
  - Israeli-Georgian Medical Research Clinic Healthycore, LTD, Tbilisi
  - LTD New Hospitals, Tbilisi
  - Pineo Medical Ecosystem, Tbilisi
  - LTD National Center of Urology Named after L. Managadze, Tbilisi
  - Multiprofile Clinic Consilium Medulla, Tbilisi
- Germany (6):
  - Friedrich Baur Institute, München, Bavaria
  - University Hospital Essen, Essen, North Rhine-Westphalia
  - Universitatsklinikum Munster, Münster, North Rhine-Westphalia
  - Universitatsklinikum Leipzig, Leipzig, Saxony
  - Charite - Universitatsmedizin Berlin, Berlin
  - Universitatsklinikum Jena, Jena
- India (14):
  - Government General Hospital, Guntur, Guntur, Andhra Pradesh
  - Institute of Neurosciences, Surat, Gujarat
  - Nizam's Institute of Medical Sciences (NIMS), Panjagutta, Hyderabad
  - Kasturba Medical College (KMC), Udupi, Karnataka
  - Amrita Institute of Medical Sciences and Research Centre (AIMS), Kochi, Kerala
  - Deenanath Mangeshkar Hospital and Research Centre, Pune, Maharashtra
  - Seth G.S. Medical College & K.E.M. Hospital, Mumbai, Pārel, Mumbai
  - All India Institute of Medical Sciences New Delhi, New Delhi, National Capital Territory of Delhi
  - Polakulath Narayanan Renai Medicity Multi Specialty Hospital, Kochi, Kochi, Punjab
  - Christian Medical College & Hospital, Ludhiana, Punjab
  - Apex Hospital, Jaipur, Rajasthan
  - City Neuro Centre, Hyderabad, Hyderabad, Telangana
  - Bangalore Medical College and Research Institute (BMCRI) - Victoria Hospital, Bangalore
  - Postgraduate Institute of Medical Education & Research, Chandigarh
- Italy (5):
  - Azienda Ospedaliera Sant'andrea, Rome, Lazio
  - Fondazione IRCCS Di Rilievo Nazionale Istituto Nazionale Neurologico Carlo Besta, Milan, Lombardy
  - Azienda Ospedaliero Universitaria Pisana, Pisa, Tuscany
  - Azienda Ospedaliera Papa Giovanni XXIII, Bergamo
  - Universita' Degli Studi di Roma La Sapienza, Roma
- Japan (12):
  - Kobe City Medical Center General Hospital, Kobe, Hyōgo
  - Kochi Medical School Hospital, Nankoku, Kochi
  - Okinawa National Hospital, Ginowan-Shi, Okinawa
  - Okinawa Prefectural Nanbu Medical Center and Children's Medical Center, Shimajiri, Okinawa
  - Saitama Medical University, Saitama Medical Center, Kawagoe, Saitama
  - Medical Hospital of Tokyo Medical and Dental University, Bunkyo, Tokyo
  - Tokyo Medical University Hospital, Shinjuku, Tokyo
  - Nihon University Itabashi Hospital, tabashi City, Tokyo
  - Yamaguchi University Hospital, Ube, Yamaguchi
  - Chiba University Hospital, Chiba
  - Hiroshima City Hiroshima Citiz, Hiroshima
  - Japanese Red Cross Osaka Hospital, Osaka
- Poland (6):
  - Clinical Research Center Spolka z Ograniczona Odpowiedzialnoscia Medic-R Sp.k, Poznan, Greater Poland Voivodeship
  - NZOZ Neuro-kard, Poznan, Greater Poland Voivodeship
  - Centrum Neurologii Klinicznej, Krakowska Akademia Neurologii, Krakow, Lesser Poland Voivodeship
  - NeuroProtect, Warsaw, Mazovian
  - Uniwersyteckie Centrum Kliniczne WUM, Centralny Szpital Kliniczny, Warsaw, Mosavian
  - Gdanski Uniwersytet Medyczny, Gdansk, Pomeranian Voivodeship
- University Clinical Centre Nis, Niš, Serbia
- South Korea (2):
  - Kyungpook National University Chilgok Hospital, Daegu
  - Samsung Medical Center, Seoul
- Spain (2):
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitari i Politecnic La Fe, Valencia
- Taiwan (5):
  - Chang Gung Memorial Foundation Kaohsiung Branch, Kaohsiung City
  - China Medical University, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Shin Kong Wu Ho Su Memorial Hospital, Taipei
  - Chang Gung Memorial Hospital at Linkou, Taoyuan District
- Turkey (Türkiye) (4):
  - Kocaeli University Hospital, Izmit, Van
  - Dokuz Eylul University Medical Faculty, Izmir
  - Ondokuz Mayis Universitesi Tip Fakultesi Hastanesi, Samsun
  - Karadeniz Technical University Farabi Hospital, Trabzon
- United Kingdom (2):
  - Sheffield Teaching Hospital NHS Foundation Trust, Sheffield, South Yorkshire
  - University Hospital Birmingham, Birmingham

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has:
  * received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication or has globally discontinued development of the product for all indications on or after April 2020 and has no plans for future development
  * made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry),
  * the legal authority to share the data, and
  * ensured the ability to protect participant privacy.
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/